CLINICAL TRIAL: NCT03301129
Title: Effects on Oxidative Stress and Platelet Activation of Traditional Cigarettes, E-cigarettes and IQOS Cigarettes: A Randomized in Vivo Study.
Brief Title: Role of Traditional Cigarettes, Electronic and IQOS Cigarettes on Oxidative Stress.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Coluzzi Flaminia (Unknown); Peruzzi Mariangela (Unknown); Nocella Cristina (Unknown); Loffredo Lorenzo (Unknown); Marullo Antonino G.M. (Unknown); Valenti Valentina (Unknown); Chimenti Isotta (Unknown); De Falco Elena (Unknown); Sciarretta Sebastiano (Unknown)
Responsible Party: Principal Investigator, Roberto Carnevale, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3241
Record Dates: First submitted 2017-09-23; First posted 2017-10-04 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Oxidative Stress Induction; Endothelial Dysfunction; Platelet Activation
MeSH Terms: interventions — Smoke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional cigarette (Experimental): smoke one Traditional cigarette (with a mean nicotine content of 0.6 mg according to package label) and in a sub-group smoke a sham cigarette (an traditional cigarette without combustion).
  Interventions: Behavioral: Smoke
- Electronic cigarette (Experimental): smoke a tobacco-flavored Electronic cigarette (9 puffs approximately equivalent to 0.6 mg of nicotine content) and in a sub-group smoke a sham cigarette (an electronic cigarette without nicotine).
  Interventions: Behavioral: Smoke
- Heat-not-burn tobacco products (IQOS) (Experimental): smoke one IQOS cigarette (with a mean nicotine content of 0.6 mg according to package label).
  Interventions: Behavioral: Smoke

INTERVENTIONS:
Behavioral: Smoke — See arm/group descriptions.

SUMMARY:
Electronic cigarettes (E-cigarettes) and new heat-not-burn tobacco products such as IQOS®, an electronic device that heats a cigarette-like stick without combustion, are a modern and technological surrogate of traditional tobacco cigarettes (T-cigarettes), that are entering in the commercial market. While the negative effects of the traditional cigarette are well known, little data are reported in scientific literature on the risks on the health by these new smoking devices. Endothelial dysfunction evaluated by flow-mediated dilatation (FMD), oxidative stress and platelet activation have been recognized as a hallmark of preclinical systemic atherosclerosis and as a useful marker to stratify the risk of cardiovascular disease in patients at risk or with established clinically significant atherosclerosis. Since no data are reported about the effects of these new smoking device on oxidative stress, platelet activation and FMD, the investigators designed a human study assessing if these new smoking devices have effects on healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* Smokers volunteers, minimum age 18 years

Exclusion Criteria:

* no history of acute or chronic organic, metabolic and inflammatory diseases;
* no fever and infections in the last 3 months;
* no history of cardiovascular pathological symptoms;
* no allergies;
* none of the participants took vitamin E, other antioxidant supplements or other drugs potentially affecting oxidative stress or FMD
* women were not menstruating when the experiment was performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
Endothelial dysfunction | up to 24 weeks
  flow-mediated dilatation (FMD) assessed by vascular ultrasound
Oxidative stress | up to 24 weeks
  Soluble Nox2-derived peptide, a direct marker of NADPH oxidase activation

SECONDARY OUTCOMES:
Platelet activation | up to 24 weeks
  evaluation of sPselectin, thromboxane and aggregation as markers of platelet activation

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Frati, MD, Study Director — Sapienza University of Rome, Policlinico Umberto I
Locations (1):
- Sapienza University, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided
identified individual participant data for all outcomes measures will be made available to other reserachers.

REFERENCES:
- [Derived] Biondi-Zoccai G, Sciarretta S, Bullen C, Nocella C, Violi F, Loffredo L, Pignatelli P, Perri L, Peruzzi M, Marullo AGM, De Falco E, Chimenti I, Cammisotto V, Valenti V, Coluzzi F, Cavarretta E, Carrizzo A, Prati F, Carnevale R, Frati G. Acute Effects of Heat-Not-Burn, Electronic Vaping, and Traditional Tobacco Combustion Cigarettes: The Sapienza University of Rome-Vascular Assessment of Proatherosclerotic Effects of Smoking ( SUR - VAPES ) 2 Randomized Trial. J Am Heart Assoc. 2019 Mar 19;8(6):e010455. doi: 10.1161/JAHA.118.010455. PMID 30879375